CLINICAL TRIAL: NCT03991299
Title: Investigating Effects of BOTOX on Weight Loss and Glucose Tolerance in Obese, Type 2 Diabetic Subjects
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Sponsor Decision.
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Naji Abumrad, John L. Sawyers Professor and Chair; Chairman Emeritus, Vanderbilt University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 181978
Record Dates: First submitted 2019-06-07; First posted 2019-06-19 (Actual); Results first posted 2023-02-28 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Obese; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2 | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Botox Arm (Experimental): Botox will be injected into duodenums of subjects via endoscopy.
  Interventions: Drug: Botox 200 UNT Injection

INTERVENTIONS:
Drug: Botox 200 UNT Injection — Botox will be injected into duodenums of subjects by endoscopy.
  Other Names: Botox

SUMMARY:
The investigators will recruit obese subjects with pre-diabetes or type 2 diabetes for the proposed clinical study for 5 visits. After informed written consent is obtained, subjects will be admitted to the Clinical Research Center, and will undergo upper endoscopic injection of Botox into the duodenal wall. The investigators anticipate that injections of Botox into the duodenal wall will result in significant weight loss and improvements in glucose tolerance and duodenal nutrient sensitivity. Subjects will be studied over a period of 6 months. Subjects will be asked to complete 5 study visits: On the first visit, each subject will undergo an oral glucose tolerance test. At visit 2, subjects will undergo an esophagogastroduodenoscopy procedure for the delivery of Botox to the duodenal wall. Visits 3-5 will be made 1, 3, and 6 months later. On every study visit, body weight and body composition will be recorded and oral glucose tolerance test will be performed. Nutrient sensing test will be performed at visits 1 and 3.

DETAILED DESCRIPTION:
Obese subjects (body mass index ≥ 30 kg/m2) with prediabetes or type 2 diabetes will be recruited by solicitation flyers, advertisements, and mass emails. Subjects who do not qualify for bariatric surgery, or subjects who are awaiting insurance approval for a bariatric procedure at the Center of Surgical Weight Loss at Vanderbilt University Medical Center will also be contacted via emails and telephone calls. Subjects will be directed to contact the researcher (Drs. Abumrad and Sundaresan) directly for more information. The recruiter will review inclusion and exclusion criteria and explain the study procedures, duration of the study and potential risks. If the subject indicates interest, screening will be performed to determine eligibility.

Subjects will undergo an initial screen by the study coordinator or research staff to assess eligibility and ability to comply with the study requirements. Prior to each study visit, subjects on oral anti-diabetic medications will be asked to discontinue these medications 4 days prior to their study visit. Diabetic subjects will be instructed to monitor their pre-prandial blood glucose during this time and to contact the study physician if their blood glucose levels are greater than 250 mg/dL for two consecutive readings. The study physician may instruct the subject to initiate short-term insulin therapy or resume their oral anti-diabetic medications; in either case the subject will be excluded from the study. Subjects will be instructed to maintain their usual diet and physical activity levels for 1 week prior to each study visit and to arrive fasted for every visit (only water after dinner).

6. Study Procedures

The subjects will be recruited for 5 study visits. After informed, written consent is obtained, subjects will be admitted to the Clinical Research Center.

Study visit 1:

Day 1:

* Subjects will arrive after an overnight fast.
* They will undergo standard physical examination; anthropometric measurements (height, weight, waist and hip circumference) perform body composition assessment via dual-energy x-ray absorptiometry imaging will be recorded.
* Baseline glucose tolerance will be assessed by an oral glucose tolerance test.
* Subjects will be handed a visual analog scale questionnaire designed to capture their perceived hunger and satiety sensations, food preferences, cravings, and feeding behavior prior to intervention. The questions will be explained by the researcher and subjects will be instructed to bring in the completed questionnaire on their second visit.
* Subjects will be provided snacks and asked to return at 7 pm for the nutrient sensing test to be performed the following day. The subject will be fed a standardized meal and restricted to water after 8:00 pm.

Day 2

* Blood will be drawn for determination of fasting plasma insulin, and gut hormones including ghrelin, Gastric inhibitory peptide, glucagon like peptide-1, pancreatic polypeptide and Peptide YY.
* Subject will then consume a standardized 250 kcal liquid mixed meal containing 40 g carbohydrates, 6 g fat, and 9 g protein within 10 minutes. Blood will be drawn at 15, 30, 60, and 120 minutes after consumption following which subject will be discharged.

Study visit 2 (within 2 weeks after the first visit):

* Subjects will undergo esophagogastroduodenoscopy procedure for the delivery of BOTOX to the duodenal wall, to be performed by Dr. Patrick Yachimski at the Vanderbilt Gastrointestinal Endoscopy Suite. The investigators have been exempted from Investigational New Drug (IND) regulation for the proposed testing by the FDA.
* Subjects will be monitored for at least two hours and discharged with instructions for follow-up and contact information of the physicians' team (Drs. Abumrad, Yachimski).

Study Visits 3-5 (1, 3, and 6 months after endoscopy): On every study visit, body weight, body composition, food intake, and feeding behavior will be recorded and post-absorptive glucose tolerance will be performed. Nutrient sensing test will be repeated at visit 3.

Oral Glucose Tolerance Test (Study visits 1 and 3-5):

* Day 0: Subjects will be fasting overnight (and restricted to water only after 8 pm).
* Day 1: Blood will be drawn for determining fasting blood glucose levels. At 8:00 am subjects will drink a solution of 75 grams dextrose in 300 ml of water in 10 minutes. Blood will be drawn at 15, 30, 45, 60, and 120 min post ingestion.
* The subject will be fed a standardized snack and discharged around noon.

Endoscopic delivery of BOTOX (Study Visit 2):

* Subjects will arrive fasted at the GI Suite in the main hospital at Vanderbilt University for the procedure.
* Under the supervision of an anesthesiologist, subjects will be given combination of intravenous medications, so they fall asleep. Dr. Yachimski will then pass the endoscope, a long, flexible tube with light, video camera and channel for small instruments including syringes through the esophagus and stomach, pylorus into the junction of the 1st and 2nd parts of the duodenum. Botox (100 units dissolved in 200 μL of sterile, preservative-free 0.9% Sodium Chloride) will be injected along the medial (mesenteric) border, into the duodenal muscle wall.

Post endoscopy Care:

* Following completion of endoscopy procedure and emergence from anesthesia, subjects will be monitored in the dedicated post-anesthesia care unit prior to discharge.
* Subjects will be provided written instructions regarding potential signs and symptoms of adverse events, including fever, pain, bleeding, and muscle weakness. They will be provided the physician call number for any questions or issues that may arise.

Nutrient sensing test (study visit 1 and 3):

* Day 1: After oral glucose tolerance test subjects return at 7:00 pm. They will be fed a standardized meal and fasted overnight (restricted to water after 8:00 pm).
* Day 2: At 8:00 am, blood will be drawn for determination of fasting plasma insulin and gut hormones stated above. Subject will then consume a standardized 250 kcal liquid mixed meal containing 40 g carbohydrates, 6 g fat, and 9 g protein to be administered over a 10-min period. Blood will be drawn 15, 30, 60, and 120 minutes later. At the end of the study, subject will be provided a standardized meal/snack and discharged.

ELIGIBILITY:
Inclusion Criteria:

1. Age = 18-65
2. BMI ≥ 30 kg/m2
3. Having established diagnosis of Type 2 diabetes or pre-diabetes

Exclusion Criteria:

1. Patients on insulin therapy
2. Endoscopy within the past 6 weeks
3. Prior bariatric surgery
4. Anti-obesity drugs
5. Serum Creatinine > 1.5 mg/dL
6. Hepatic enzyme elevations > 2x the upper limits of normal
7. Current use of warfarin
8. Abnormal ECG
9. Positive pregnancy test for female subjects in the child bearing age
10. Pre-existing cardiovascular disease (heart attack in the past 3 months, cardiac stenting, heart valve disorders)
11. Prior surgery on the alimentary tract
12. Gastroparesis
13. Inflammatory bowel disease
14. Liver failure

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2021-04-29 (Actual); Primary Completion 2022-02-11 (Actual); Study Completion 2022-02-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Naji Abumrad, MD, Study Director — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 4 participants enrolled.
  1 participants withdrew.
Period: Overall Study
Arm/Group | Botox Arm
Started | 4
Completed | 0
Not Completed | 4
Not completed — Study closed, sponsor decision | 3
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: Participants analysis not done.
Arm/Group | BOTOX Arm
Number analyzed (Participants) | 4
Age, Continuous [Mean (Full Range); unit: years] | 43.7 [21.7 to 56.1]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Body Weight at 6 Months
Description: Body weight will be measured at baseline and 6 months after Botox injections.
Time Frame: Baseline - 6 months
Population: Data analysis could not be completed as zero participants remained enrolled in the study for 30 days or more
Arm/Group | Botox Arm
Number analyzed (Participants) | 0

2. Primary Outcome: Change in Body Weight at 3 Months
Description: Body weight will be measured at baseline and 3 months after Botox injections.
Time Frame: Baseline - 3 months
Population: Data analysis could not be completed as zero participants remained enrolled in the study for 30 days or more
Arm/Group | Botox Arm
Number analyzed (Participants) | 0

3. Primary Outcome: Change in Body Weight at 1 Month
Description: Body weight will be measured at baseline and 1 month after Botox injections.
Time Frame: Baseline - 1 month
Population: Data analysis could not be completed as zero participants remained enrolled in the study for 30 days or more
Arm/Group | Botox Arm
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Baseline to four weeks
Arm/Group | Botox Arm
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 1/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Botox Arm (N=4)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) — MH02 - Abdominal pain (6.5/10) the night of EGD - intermittent but frequent
Joint pain (Musculoskeletal and connective tissue disorders) | 1 (1) — Left rib facet pain and inflammation.

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects enrolled.

Technical problems due to limited enrollment leading to uninterpretable data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-08): https://cdn.clinicaltrials.gov/large-docs/99/NCT03991299/Prot_SAP_000.pdf